CLINICAL TRIAL: NCT03299530
Title: Accuracy of Corneal Astigmatism in Different Region Modes
Status: Recruiting | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, A-Yong Yu, Director of the Cataract Clinical Center, Wenzhou Medical University
Other Study IDs: 2017ASTIGMATISM REGIONS
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Astigmatism; Cornea
Keywords: Corneal Astigmatism; Scheimpflug; pupil size; Toric
MeSH Terms: conditions — Astigmatism; Corneal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with corneal astigmatism: Patients who had received phacoemulsification surgery with or without implantation of toric IOL are with a certain amount of corneal astigmatism.
  Interventions: Other: patients with corneal astigmatism

INTERVENTIONS:
Other: patients with corneal astigmatism — The total corneal astigmatism, anterior chamber depth, will be measured by a Scheimpflug tomographer. Pupil size will be measured by itrace device and MONCV3 device. Residual astigmatism will be tested by subjective refraction.

SUMMARY:
To analyze the difference between measured total corneal astigmatism and actual corneal astigmatism under different region modes and optimize the region setting.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients who had received phacoemulsification surgery with or without implantation of toric IOL are with a certain amount of corneal astigmatism.
* Best corrected visual acuity ≥ 0.66 (20/30 Snellen)

Exclusion Criteria:

* Corneal diseases or severe irregular astigmatism (e.g., pterygium, keratoconus), existence of corneal opacification;
* Ocular disease which may affect visual acuity (e.g., glaucoma, uveitis, retinal disease, pathologic myopia);
* History of ocular surgery or ocular trauma before this cataract surgery;
* Decentration of IOL > 0.3mm or tilt > 5°
* Implantation of multifocal IOL
* history of wearing of rigid contact lens within the past 4 weeks or soft contact lens within 1 week;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received cataract surgery in The Eye Hospital of Wenzhou Medical University
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-10-28 (Estimated)

PRIMARY OUTCOMES:
Vectorial difference | ≥1 month after surgery
  The vectorial difference between measured corneal astigmatism (under multiple different region mode settings) and actual corneal astigmatism.
pupil size | ≥1 month after surgery
  pupil size of patients in a bright environment measured by itrace device and MONCV3 device
pupil size 2 | ≥1 month after surgery
  pupil size of patients measured by Pentacam HR device
residual astigmatism | ≥1 month after surgery
  residual astigmatism tested by subjective refraction
total corneal astigmatism | ≥1 month after surgery
  Total corneal astigmatism measured by a scheimpflug tomographer under different region mode settings.
Anterior chamber depth | ≥1 month after surgery
  The distance between corneal apex and anterior surface of IOL measured by a scheimpflug tomographer
actual corneal astigmatism | ≥1 month after surgery
  actual corneal astigmatism is derived from residual astigmatism at corneal plane and cylindrical power of IOL at corneal plane through Holladay 2 formula.

CONTACTS AND LOCATIONS:
Overall Officials: AYong Yu, MD.PhD., Principal Investigator — Wenzhou Medical University
Locations (1):
- Eye Hispital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No